CLINICAL TRIAL: NCT04679467
Title: An Acceptability Study to Evaluate the Tolerance, Adherence and Metabolic Control of Patients With Phenylketonuria (PKU) Consuming PKU Sphere™, a Glycomacropeptide (GMP) Based Protein Substitute, When Introduced According to a Practical Guide to PKU Sphere.
Brief Title: Evaluation of PKU Sphere in Italy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT-W-GMPIT-2019-03-08
Record Dates: First submitted 2020-11-26; First posted 2020-12-22 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonurias; PKU
Keywords: Phenylketonuria; PKU; Glycomacropeptide; Food for Special Medical Purposes
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Open-label, single group interventional study.
Masking Description: Open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental - single arm (Experimental): All patients to recieve PKU sphere as part of their dietary management for phenylketonuria (PKU)
  Interventions: Dietary Supplement: PKU sphere

INTERVENTIONS:
Dietary Supplement: PKU sphere — TYR sphere is a powdered, low phenylalanine and tyrosine protein substitute, containing a balanced mix of casein glycomacropeptide (cGMP) isolate, essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals and the long chain polyunsaturated fatty acid (LCP); Docosahexaenoic acid (DHA). It contains sugars and sweetener.
  The product is designed to be prescribed based on its protein content, not its energy content.

SUMMARY:
20 participants with PKU will build-up their dietary intake of PKU sphere over 2-16 weeks, depending on their level of metabolic control whilst doing so. Participants will complete a gastrointestinal specific and PKU specific questionnaire at the Baseline clinic visit and record the amount of PKU sphere taken each day. Dried blood spots are taken twice per week.

Once built up to a clinically appropriate intake of PKU sphere, or after 16 weeks, participants enter a 4-week Evaluation Period. The amount of PKU sphere taken per day continues to be recorded by participants. Gastrointestinal tolerance over the preceding seven days is recorded at the end of each week. Evaluations of PKU sphere's palatability are made at the end of weeks two and four of the Evaluation Period. Dried blood spots are taken once per week.

The participant attends an End of Study Visit at the clinic and the investigator decides whether they should continue taking PKU sphere.

DETAILED DESCRIPTION:
20 participants with phenylketonuria (PKU) will introduce PKU sphere into their diet. PKU sphere is a food for special medical purposes (as defined by Regulation (EU) No 609/2013 on food for specific groups), used for the dietary management of phenylketonuria from 3 years of age.

The study begins with a Baseline clinic visit. Informed consent is taken by the investigator before the participant completes a PKU specific quality of life questionnaire, and a GI specific questionnaire. The participant takes a dried blood spot in order for the investigator to check their technique is correct.

Build-up and Stabilisation Period. This will last between 2 and 16 weeks, depending on how long the participant takes to reach their maximum recommended intake of PKU sphere. Participants will take a dried blood spot twice per week in order for their health care professional to monitor their phenylalanine and tyrosine levels. After three consecutive dried blood spot results within the target range, the participant's HCP can advise to swap one portion of amino acid-based protein substitute for PKU sphere. This method of building up the amount of PKU sphere to be taken is informed directly by Vitaflo's 'Practical Guide to PKU sphere'. The amount of PKU sphere taken each day is recorded by the participant in their study diary.

Once the maximum recommended amount of PKU sphere is being taken by the participant, or after 16 weeks, the participant moves into the four-week Evaluation Period. Participants then take a dried blood spot once per week, but continue to record their intake of PKU sphere each day. At the end of each Evaluation Period week, participants record any gastrointestinal symptoms experienced over the preceding seven days. At the end of Evaluation Period weeks two and four, participants will also record their thoughts on PKU sphere's palatability. This includes a Likert scale rating of the product's appearance, taste, aftertaste, smell, texture, packaging and ease of use.

At the end of the Evaluation Period, participants return to the clinic for the End of Study visit. The PKU and GI specific questionnaires completed at Baseline are repeated and the Investigator discusses the suitability of the participant to continue to take PKU sphere as part of their regular therapeutic diet. Following the visit, the Investigator rates the utility of the Practical Guide to PKU sphere. A Follow-up Phone Call will relay the results of any outstanding dried blood spot results to participants following their End of Study Visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PKU or hyperphenylalaninemia via new born screening and early treated, requiring >50% of protein intake from protein substitute.
* Aged 3 years and above.
* Female patients of childbearing potential must have a negative urine pregnancy test prior to completing the screening procedures.
* Willingly given, written, informed consent from the participant, 18 or more years, or from the parent/guardian for participants < 18 years.
* Willingly given, written assent (if appropriate) for those < 18 years.

Exclusion Criteria:

* Pregnant, planning pregnancy or breastfeeding.
* Intake of sapropterin dihydrochloride (Kuvan), PEG PAL or large neutral amino acids within 30 days prior to screening visit.
* Patients currently taking their maximum recommended amount of protein substitute from a GMP based protein substitute.
* Patients who are unable/unwilling to replace their current GMP protein substitute (if any) with PKU sphere.
* Patients with known soya, milk or fish allergies / intolerance.
* Individuals, who in the opinion of the investigator, are unable to comply with the requirements of the protocol.
* Any co-morbidity, which in the opinion of the Investigator, would preclude participation in the study.
* Patients who are currently participating in, plan to participate in, or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to screening visit.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in adherence to recomended amounts of PKU sphere | Recorded daily from start of 2-16 week Build-up and Stabilisation Period to end of 4 week Evaluation Period, assessed by HCPs periodically as per routine practice.
  Patient reported data on actual compared to prescribed intakes of PKU sphere
Change in gastrointestinal tolerance | Data on previous 7 days collected by patients at the end of each Evaluation Period week. This data will be assessed by HCPs periodically as per routine practice.
  Patient reported data on any gastrointestinal symptoms experienced
Patient evaluation of PKU sphere's palatability, Evaluation Period week 2 | End of Evaluation Period week 2.
  Patient reported Likert-scale evaluation of PKU sphere's appearance, smell, taste, aftertaste, texture, packaging/presentation and ease of use. A higher score denotes a more positive response.
Patient evaluation of PKU sphere's palatability, Evaluation Period week 4 | End of Evaluation Period week 4.
  Patient reported Likert-scale evaluation of PKU sphere's appearance, smell, taste, aftertaste, texture, packaging/presentation and ease of use. A higher score denotes a more positive response.
Change in metabolic control (phenylalanine) over Build-up and Stabilisation Period. | Dried blood spots taken twice weekly during 2-16 week Build-up and Stabilisation Period.
  Phenylalanine levels obtained from dried blood spots
Change in metabolic control (phenylalanine) over Evaluation Period. | Dried blood spots taken once weekly during 4-week Evaluation Period.
  Phenylalanine levels obtained from dried blood spots
Change in metabolic control (tyrosine) over Build-up and Stabilisation Period. | Dried blood spots taken twice weekly during 2-16 week Build-up and Stabilisation Period.
  Tyrosine levels obtained from dried blood spots
Change in metabolic control (tyrosine) over Evalaution Period. | Dried blood spots taken once weekly during 4-week Evalaution Period.
  Tyrosine levels obtained from dried blood spots
Change in gatrointestinal quality of life | Baseline visit (day one) and End of Study visit (post day-28 of Evaluation Period)
  Age-specific, GI related quality of life questionnaire completed by participants. The specific version of the questionnaire to be used by each age group is listed below:
  Age 2-4 years (Parental completion) = MAPI PedsQL Gastrointestinal Symptoms Scales, Toddlers (2-4) Age 5-7 years (Parental completion) = MAPI PedsQL Gastrointestinal Symptoms Scales, Young Children (5-7) Age 8-12 years (Parental completion) = MAPI PedsQL Gastrointestinal Symptoms Scales, Children (8-12) Age 13-18 years = MAPI PedsQL Gastrointestinal Symptoms Scales, Teens (13-18) Age 18 years and upwards = Birmingham IBS Symptom Questionnaire
  The MAPI PedsQL Gastrointestinal Symptoms Scale questionnaires and the Birmingham IBS symptom Questionnaire indicate fewer problems with higher calculated scores.
Change in PKU specific quality of life | Baseline visit (day one) and End of Study visit (post day-28 of Evaluation Period)
  Age-specific, PKU related quality of life questionnaire completed by participants. The specific version of the questionnaire to be used by each age group is listed below:
  Age >9 years = MAPI phenylketonuria impact and treatment Quality Of Life Questionnaire (PKU-QOL), Parents Age 9-11 years = MAPI phenylketonuria impact and treatment Quality Of Life Questionnaire (PKU-QOL), Children Age 12-17 years = MAPI phenylketonuria impact and treatment Quality Of Life Questionnaire (PKU-QOL), Adolescent Age 18+ years = MAPI phenylketonuria impact and treatment Quality Of Life Questionnaire (PKU-QOL), Adult
  With all versions of the PKU-QOL, a higher calculated score denotes higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Marchesini Reggiani, Principal Investigator — Universita di Bologna
Locations (4):
- Italy (4):
  - Sant'Orsola-Malpighi Polyclinic (adults), Bologna
  - Sant'Orsola-Malpighi Polyclinic (paediatrics), Bologna
  - Ospedale San Paolo, Milan
  - A.O.R.N. Santobono-Pausilipon - Ospedale Santobono, Napoli

IPD SHARING:
Plan to Share IPD: No